CLINICAL TRIAL: NCT03438578
Title: Use of Efficacy Safety Score in Postoperative Management: A Prospective, Randomized Study
Brief Title: Efficacy Safety Score in Postoperative Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/1903
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
Keywords: Patient safety; Postoperative care; Monitoring, physiologic; Safety management
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy Safety Score monitoring (Experimental): Patients monitored with wireless vital signs and Efficacy Safety Score after discharge from the post-anesthesia care unit to an ordinary ward
  Interventions: Device: Efficacy Safety Score monitoring
- Regular (No Intervention): Patients receiving standard postoperative care after discharge from the post-anesthesia care unit to an ordinary ward

INTERVENTIONS:
Device: Efficacy Safety Score monitoring — According to data gathered from ESS and monitoring, the patients will receive needed care.
  Other Names: Isansys, Patient Gateway System
  Arms: Efficacy Safety Score monitoring

SUMMARY:
The primary aim of this project is to determine whether postoperative patients may benefit from the Efficacy Safety Score (ESS) as a tool for postoperative clinical decision support, with a special focus on the first 24 hours after discharge from the postoperative care unit.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery
* expectedly to be treated and observed in hospital for more than 24 hours postoperatively

Exclusion Criteria:

* refusal of participation
* poor communication capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Raeder, Prof, Study Director — University of Oslo; Erik Solligård, MD PhD, Study Director — St. Olavs Hospital
Locations (1):
- St Olav University Hospital, Orkdal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Skraastad EJ, Borchgrevink PC, Nilsen TIL, Raeder J. Postoperative quality and safety using Efficacy Safety Score (ESS) and a wireless patient monitoring system at the ward: A randomised controlled study. Acta Anaesthesiol Scand. 2020 Mar;64(3):301-308. doi: 10.1111/aas.13492. Epub 2019 Nov 12. PMID 31608431

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efficacy Safety Score Monitoring | Regular
Started | 100 | 100
Completed | 99 | 96
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efficacy Safety Score Monitoring | Regular | Total
Number analyzed (Participants) | 96 | 99 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] — Patients > 18 years of age undergoing acute or elective surgery expected to be hospitalised > 24 hours postoperatively.
  Years | 61 (12.5) | 62 (13.3) | 62 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 60 | 62 | 122
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Norway | 96 | 99 | 195

OUTCOME MEASURES:

1. Primary Outcome: Time to Mobilization
Description: The measured postoperative time when patient can stand and able to walk one or more steps, with or without support
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Efficacy Safety Score Monitoring | Regular
Number analyzed (Participants) | 96 | 99
hours | 10.1 [8.1 to 12.2] | 14.2 [12.0 to 16.3]

2. Secondary Outcome: Pain Measurement, Verbal Numeric Rating Scale
Description: Reported pain hourly on a 11-digit scale, called Verbal Numeric Rating Scale for pain, 0-10 where 0 is no pain, and 10 is worst thinkable pain. Higher scores mean a worse outcome.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Efficacy Safety Score Monitoring | Regular
Number analyzed (Participants) | 96 | 99
score on a scale | 2.1 [1.8 to 2.9] | 3.3 [2.9 to 3.7]

3. Secondary Outcome: Patient Satisfaction
Description: Reported patient satisfaction on a 1-5 scale, (Likert scale), where 1 is Very dissatisfied, and 5 is Very satisfied. Higher scores mean a better outcome.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Efficacy Safety Score Monitoring | Regular
Number analyzed (Participants) | 96 | 99
score on a scale | 4.9 [4.9 to 5.0] | 4.3 [4.2 to 4.5]

ADVERSE EVENTS:
Time Frame: 24 hour after surgery
Description: Low blood pressure Arrythmia Need for extra treatment Neurological events
Arm/Group | Efficacy Safety Score Monitoring | Regular
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/96 | 2/99
Other Adverse Events (participants affected / at risk) | 5/96 | 0/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efficacy Safety Score Monitoring (N=96) | Regular (N=99)
Neurological seizure (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efficacy Safety Score Monitoring (N=96) | Regular (N=99)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Pain treatment, nerve blocks (Nervous system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT03438578/Prot_SAP_000.pdf